CLINICAL TRIAL: NCT04195737
Title: Comparative Evaluation of Coronally Advanced Root Coverage Procedure With Ossix Volumax™ Collagen Matrix and Connective Tissue Graft-Randomized Controlled Trial
Brief Title: Comparison of Coronally Advanced Root Coverage Procedure With Collagen Matrix and Connective Tissue Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_100209
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Gingival Recession
Keywords: Gingival Recession Coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Two groups were made one test and control. The test group will be treated with coronally advanced flap with ossix volumax™ collagen matrix and control group will be treated with coronally advanced flap with Sub epitheial Connective Tissue Graft.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root coverage with ossix volumax collagen matrix (Experimental): Evaluation of root coverage achieved by collagen matrix in conjunction with coronally advanced flap in patients with multiple gingival recession.
  Interventions: Procedure: Ossix volumax collagen matrix
- Root coverage with connective tissue graft (Active Comparator): Evaluation of root coverage achieved by connective tissue graft in conjunction with coronally advanced flap in patients with multiple gingival recession
  Interventions: Procedure: Connective Tissue Graft

INTERVENTIONS:
Procedure: Ossix volumax collagen matrix — Under LA horizontal incision is made.Split-full-split thickness flap is elevated.The remaining soft tissue of the anatomic interdental papillae deepithelialized.Coronal advancement of the flap obtained and closed using sling suture.
  Arms: Root coverage with ossix volumax collagen matrix
Procedure: Connective Tissue Graft — Under LA parallel incisions is made 1-2 mm first molar to canine.Graft incision 1 mm coronal to the horizontal flap incision.Through this incision designed graft thickness is obtained.The graft obtained between the two horizontal incisions has a 1 mm coronal strip that require depithelisation with a knife and closed using interrupted suture.
  Arms: Root coverage with connective tissue graft

SUMMARY:
The present study is a human, prospective, randomised controlled clinical trial conducted to explore the outcome of a coronally advanced flap with ossix volumaxTM collagen matrix and connective tissue graft in the treatment of multiple adjacent gingival recession defects.

The trial is in accordance with the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
Periodontal plastic surgery are surgical procedures performed to prevent or correct anatomic, developmental, traumatic or disease-induced defects of the gingiva, alveolar mucosa or bone. It includes various soft and hard tissue procedures aimed at gingival augmentation, root coverage, correction of mucosal defects at implants, crown lengthening, gingival preservation at ectopic tooth eruption, removal of aberrant frena, prevention of ridge collapse associated with tooth extraction and augmentation of the edentulous ridge.1

Different predisposing anatomic features can result in recession such as position and anatomy of teeth in the dental arch, bony dehiscence, thickness of the alveolar mucosa, muscle pull, orthodontic treatment, thin gingival biotype, buccal prominence of teeth, lack of keratinized tissue, abnormal frenum attachment, or patient related factors such as vigorous brushing or chronic gingival inflammation.2 The migration of the marginal tissue to an apical position may lead to esthetic concern, dentin hypersensitivity, root caries, and cervical wear. Treatment modalities for gingival recession have many influencing factors such as defect dimensions (depth, width), site (maxilla, mandible), defect number (single, multiple), soft tissue anatomy (keratinized tissue quality/quantity; papilla height/width; frenum/ muscle pull; vestibular depth) tooth position etc.

Various surgical techniques for the treatment of recessions includes the use of full or partial thickness flap with various soft tissue grafts such as epithelized free gingival grafts (FGG) or sub-epithelial connective tissue graft (SCTG) in conjunction with various types of flaps eg: (envelope, coronally or laterally positioned flap, double pedicle flap (DPF) or tunnelling (TUN) alone or combined with laterally positioned pedicle flaps (LPPF).3 Coronally advanced flap (CAF) with connective tissue graft (CTG) is considered as the gold standard treatment for gingival recession. Commercially available materials for root coverage are expanded Poly Tetra Fluoro Ethylene (Gore-Tex), polglactin, Collagen membranes like biogide, biomend, resolute, alloderm, collatape etc, collagen matrix such as mucograft, human amniotic membrane, dermagraft, ossix.4

Recently in a case report using platelet concentrate carried on collagen sponge (ossix) showed favourable results.4 Ossix volumax™ has shown De novo bone formation when used in alveolar ridge augmentation procedure.5

Ossix volumax™ (Datum dental) is one such recently identified sugar cross-linked bio programmed collagen matrix. Ossix volumax™ is a volumizing, thick collagen scaffold, featuring glymatrix technology. The properties are thick and expand when wet, excellent handling, easy to use, adapts and adheres to the bone.5 It undergoes rapid ossification (in CT scans and histology after one month).6

Literature search till date has shown no studies regarding the use of type 1 sugar cross-linked collagen membrane for treatment of gingival recession. So, the present study is undertaken with the aim to comparatively evaluate the advantages of ossix volumax collagen membrane with subepithelial connective tissue graft for the treatment of multiple adjacent gingival recession defects.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to18 years.
* Multiple adjacent Miller's class I and class II gingival recession sites.
* Patients with healthy or treated periodontal conditions.
* Patients with esthetic concerns.
* Absence of uncontrolled medical conditions.
* Full mouth plaque score </= 10% (O'Leary 1972)
* Full mouth bleeding score <10% (Ainamo and Bay 1975)

Exclusion Criteria:

* Gingival biotype less than 0.8 mm.
* Pregnant or lactating females.
* Tobacco smoking.
* Untreated periodontal conditions.
* Use of systemic antibiotics in the past 3 months.
* Patients treated with any medication known to cause gingival hyperplasia

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
gingival recession depth | 6 months
  measured as the distance from the CEJ to the gingival margin.
Complete root coverage | 6 months
  root coverage regarded as complete with gingival margin located at the level of Cemento Enamel Junction
Mean root coverage | 6 months
  (Baseline recession depth - 6 month recession depth/Baseline recession depth)*100

SECONDARY OUTCOMES:
pocket Probing depth | 6 months
  measured as the distance from the gingival margin to the base of gingival sulcus
Gingival Recession width | 6 months
  measured as the distance between the mesial gingival margin and distal gingival margin (measurement will be recorded on a horizontal line tangential to the cementoenamel junction).
Clinical attachment level | 6 months
  measured as Gingival Recession Depth + Probing Depth
Gingival biotype thickness | 6 months
  measured 3mm apically from the free gingival margin at the mid buccal aspect of the tooth.
Apico-coronal width of keratinized tissue | 6 months
  ) measured as the distance from the mucogingival junction to the gingival margin,with the mucogingival junction location determined using (Schiller's Potassium Iodide Solution).
Root coverage esthetic score | 6 months
  The Aesthetic evaluation was performed according to the root coverage aesthetic score system (RES).
  Five Variables evaluated which are as follows:
  Level of Gingival margin (GM) Marginal Tissue Contour (MTC) Soft Tissue Texture (STT) Mucogingival Junction(MJ) alignment Gingival Colour (GC) The values ranges between 0 - 6.Higher the value better is the outcome.
Plaque index | 6 months
  It is measured by using UNC 15 probe.The values lie between 0 - 3.Higher the outcome the prognosis will be poor.
Gingival index | 6 months
  It is measured by using UNC 15 probe.The values lie between 0 - 3.Higher the outcome the prognosis will be poor.
Gingival Bleeding index | 6 months
  It is measured by using UNC 15 probe.The values lie between 0 - 1. And presence or absence of bleeding is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Prabhuji MLV, Study Director — Krishnadevarya Dental College
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India